CLINICAL TRIAL: NCT03675555
Title: Prophylactic Mirtazapine or Dexamethasone for Post-spinal Anesthesia Shivering in Patients Undergoing Gynecological Surgeries: a Randomized Controlled Trial
Brief Title: Prophylactic Mirtazapine or Dexamethasone for Post-spinal Anesthesia Shivering
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dr.Ibrahim Mamdouh Esmat, Assistant Professor of Anesthesia and Intensive Care Department, Faculty of Medicine, Ain- shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R 47 / 2018
Record Dates: First submitted 2018-09-14; First posted 2018-09-18 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Shivering
MeSH Terms: interventions — Mirtazapine; dexamethasone 21-phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- M (Mirtazapine) (Merta) group:(n=100) (Active Comparator)
  Interventions: Drug: Mirtazapine
- D (Dexamethasone) (Dex) group: (n=100) (Active Comparator)
  Interventions: Drug: Dexamethasone phosphate
- C (Control) group: (n=100) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mirtazapine — Each patient received 30 mg Mirta tablet orally with sips of water and 100 ml 0.9% sodium chloride (normal saline [NS]) (IVI) over 15 minutes as a placebo for Dex solution 2 hours preoperatively.
  Other Names: Remeron
  Arms: M (Mirtazapine) (Merta) group:(n=100)
Drug: Dexamethasone phosphate — Each patient received a placebo tablet identical to Mirta tablet orally with sips of water and Dex 8 mg ampoule diluted in 100 ml 0.9% NS IVI over 15 minutes, 2 hours preoperatively.
  Arms: D (Dexamethasone) (Dex) group: (n=100)
Drug: Placebo — Each patient received a placebo tablet identical to Mirta tablet orally with sips of water and 100 ml 0.9% NS IVI over 15 minutes as a placebo for Dex solution 2 h preoperatively.preoperatively.
  Arms: C (Control) group: (n=100)

SUMMARY:
This study was conducted to evaluate the effect of a prophylactic dose of oral mirtazapine on shivering compared with prophylactic intravenous infusion (IVI) dexamethasone in patients undergoing gynecological surgeries under spinal anesthesia.

DETAILED DESCRIPTION:
Enrollment After approval by the institute ethics committee, this study was conducted at Ain-Shams university hospitals, from the 1st of March 2018 till the 31st of August 2018, on 300 patients aged 18-60 years of the American Society of Anesthesiologists (ASA) physical status I or II and underwent gynecological surgeries under spinal anesthesia. A written informed consent was obtained from all patients to participate in the study.

Patient's refusal, duration of surgery more than 120 min, obesity with body mass index (BMI) >35 kg/m2, generalized infection or localized infection at level of blockade, neurologic disease, coagulation disorder, patients with hypo- or hyperthyroidism, cardiopulmonary disease, psychological disorders, a need for blood transfusion during surgery, an initial body temperature >38.0C or <36.0C, a known history of alcohol or substance abuse, or receiving vasodilators, or medications likely to alter thermoregulation excluded the patient from the study.

Randomization and Blinding This study was designed to be a randomized, placebo-controlled, double-blinded parallel study. Following enrollment, patients were randomized into 3 equal groups;

1. The M (Mirtazapine) (Merta) group:(n=100) each patient received 30 mg Mirta tablet orally with sips of water and 100 ml 0.9% sodium chloride (normal saline [NS]) (IVI) over 15 min as a placebo for Dex 2 h preoperatively.
2. The D (Dexamethasone) (Dex) group: (n=100) each patient received a placebo tablet identical to Mirta tablet orally with sips of water and Dex 8 mg ampoule diluted in 100 ml 0.9% NS IVI over 15 min, 2 h preoperatively.
3. The C (Control) group: (n=100) each patient received the same placebo tablet identical to Mirta tablet orally with sips of water and 100 ml 0.9% NS IVI over 15 minas a placebo for Dex 2 h preoperatively.

Randomization was done using computer-generated table of random numbers in a 1:1 ratio in opaque and sealed envelope (SNOSE). The assigned treatment was written on a card and sealed in opaque envelopes consecutively numbered. These envelopes were opened just immediately before infusing the medication in the patient's room. The study drugs were prepared by the hospital pharmacy and follow-up of patients were conducted by anesthesia residents not involved in any other part of the study.

Study Protocol On arrival in the operating theatre, all patients had an inserted venous cannula. I.V. fluids were preheated to 37oC. No other warming device was used. Lactated Ringer's solution was warmed to 37 oC and was infused at 10 ml/kg over 30 min before spinal anesthesia. The infusion rate was reduced to 6 ml/ kg.

Subarachnoid anesthesia was instituted at either L3/4 or L4/5 interspaces. Hyperbaric bupivacaine, 5 mg /ml, 15 mg was injected using a 25 G Quincke spinal needle.

Supplemental oxygen (5 liter/ min) was delivered via a facemask during the operation. All patients were covered with one layer of surgical drapes over the chest, thighs, and calves during the operation and one cotton blanket over the entire body after operation. The operating and recovery rooms temperatures were maintained at 23-25°C with approximately 60% humidity.

Assessment parameters Heart rate, mean arterial pressure (MAP), and peripheral oxygen saturation were recorded using standard noninvasive monitors before intrathecal injection and thereafter at 5, 10, 15, 20 minutes then every 10 minutes to complete 90 minutes from the intrathecal injection.

Sensory levels were assessed by pinprick to determine the peak sensory level and time to two segment regression in minutes. Motor block were assessed by using Modified Bromage scale(16) (0 = no block 1 = hip block, 2 = hip and knee block, 3 = hip, knee, and ankle block) to determine the time to reach complete motor block and duration of motor blockade (minutes).

Sedation score was assessed with a four-point scale as per Filos et al.(17): 1: Awake and alert. 2: Somnolent, but responsive to verbal stimuli. 3: Somnolent, arousable to physical stimuli. 4: Unarousable.

Body temperature (axillary temperature) was recorded with an axillary thermometer. The ambient temperature was measured by a wall thermometer. The ambient temperature will be maintained at 25oC with constant humidity.

Shivering severity was assessed with a four-point scale (Badjatia et al):

1. None (Grade 0): no shivering noted on palpation of the masseter, neck, or chest wall
2. Mild (Grade 1): shivering localized to the neck and/or thorax only
3. Moderate (Grade 2): shivering involved gross movement of the upper extremities (in addition to neck and thorax)
4. Severe (Grade 3): shivering involved gross movements of the trunk and upper and lower extremities.

Shivering was assessed immediately before the block and every 10 minutes till the first 90 min (end point of the study) after the completion of the subarachnoid drug injection (start point of the study). Grade 2 or 3 of shivering score was regarded failure of prophylaxis and meperidine 25 mg IV was administered.

Side-effects, including hypotension (defined as a decrease in MAP of more than 20% from baseline or a decrease of arterial blood pressure below 90 mmHg and baseline MAP was calculated from three measurements taken on the ward before surgery) was treated by crystalloid infusion and if necessary ephedrine 5 mg IV was administered. The amount of ephedrine given in each group was recorded. Bradycardia was considered if the heart rate <50 beats/min and was treated with IV atropine (0.01mg/kg). Respiratory depression (RR < 12 bpm), incidence of nausea and vomiting during early 2 hours postoperatively were recorded. IV granisetron (1 mg) was given in case of vomiting or after 2 successive episodes of nausea.

Patients' satisfaction with shivering prophylaxis was done by asking the patient to answer the question, "How would you rate your experience after the surgery?" using a 7-point Likert verbal rating scale and acceptable satisfaction score of the patient being 5-7.

3-Analysis of Data:

The collected data were coded, tabulated, and statistically analyzed using IBM SPSS statistics (Statistical Package for Social Sciences) software version 22.0, IBM Corp., Chicago, USA, 2013.

ELIGIBILITY:
Inclusion Criteria:

* on 300 patients aged 18-60 years
* of the American Society of Anesthesiologists (ASA) physical status I or II
* and underwent gynecological surgeries under spinal anesthesia.
* A written informed consent was obtained from all patients to participate in the study.

Exclusion Criteria:

* Patient's refusal,
* duration of surgery more than 120 min,
* obesity with body mass index (BMI) >35 kg/m2,
* generalized infection or localized infection at level of blockade,
* neurologic disease,
* coagulation disorder,
* patients with hypo- or hyperthyroidism,
* cardiopulmonary disease,
* psychological disorders,
* a need for blood transfusion during surgery,
* an initial body temperature >38.0C or <36.0C,
* a known history of alcohol or substance abuse,
* or receiving vasodilators, or medications likely to alter thermoregulation

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
The incidence of clinically significant PSAS which required IV pethidine for treatment (Grade 2 (moderate) and Grade 3 (severe)) | The first 90 min (end point of the study) after the completion of the subarachnoid drug injection (start point of the study).
  The incidence of clinically significant PSAS which required IV pethidine for treatment (Grade 2 (moderate) and Grade 3 (severe)) after the first 90 min (end point of the study) after the completion of the subarachnoid drug injection (start point of the study).

CONTACTS AND LOCATIONS:
Locations (1):
- Ibrahim Mamdouh Esmat, Heliopolis, Cairo Governorate, Egypt

REFERENCES:
- [Derived] Esmat IM, Elsayed AM, El-Hariri HM, Ashoor TM. A Randomized Controlled Trial for Prevention of Postspinal Anesthesia Shivering in Gynecological Surgeries: Mirtazapine vs. Dexamethasone. Anesthesiol Res Pract. 2022 Mar 9;2022:5061803. doi: 10.1155/2022/5061803. eCollection 2022. PMID 35310422